CLINICAL TRIAL: NCT01157897
Title: Phase 1/2a Open-label Dose Safety, Reactogenicity, Immunogenicity and Efficacy of the Candidate Plasmodium Vivax Malaria Protein 001 (VMP001) Administered Intramuscularly With GlaxoSmithKline (GSK) Biologicals' Adjuvant System AS01B in Healthy Malaria-Naïve Adults
Brief Title: Study of VMP001 and AS01B (Adjuvant Formulation) in Healthy Malaria-Naïve Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: The PATH Malaria Vaccine Initiative (MVI) (Other); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WRAIR 1692; IND 14380 (Other: FDA)
Record Dates: First submitted 2010-07-02; First posted 2010-07-07 (Estimated); Results first posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Malaria; Plasmodium Vivax
Keywords: Malaria; Plasmodium Vivax; Vaccine
MeSH Terms: conditions — Malaria; Malaria, Vivax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1: 15 μg VMP001 (Experimental): 15ug VMP001 per vaccination on days -1 or 0, 28, and 84. P. vivax sporozoite challenge on day 98.
  Interventions: Biological: VMP001; Other: P. vivax sporozoite challenge
- Cohort 2: 30 μg VMP001 (Experimental): 30ug VMP001 per vaccination on days 14, 42, and 84. P. vivax sporozoite challenge on day 98.
  Interventions: Biological: VMP001; Other: P. vivax sporozoite challenge
- Cohort 3: 60 μg VMP001 (Experimental): 60ug VMP001 per vaccination on days 28, 56, and 84. P. vivax sporozoite challenge on day 98.
  Interventions: Biological: VMP001; Other: P. vivax sporozoite challenge
- Control (Other): No Vaccinations given for controls. P. vivax sporozoite challenge on day 98.
  Interventions: Other: P. vivax sporozoite challenge

INTERVENTIONS:
Biological: VMP001 — Plasmodium vivax malaria protein 001 (VMP001) with GSK Biologicals' Adjuvant System AS01B
  Arms: Cohort 1: 15 μg VMP001; Cohort 2: 30 μg VMP001; Cohort 3: 60 μg VMP001
Other: P. vivax sporozoite challenge — P. vivax sporozoite challenge

SUMMARY:
This is a first-in-humans safety, immunogenicity and efficacy study with recombinant protein VMP001, a Plasmodium vivax circumsporozoite (CS) protein based vaccine. This open label study will be performed in malaria-naïve adults in the United States. Three doses of VMP001 formulated in AS01B (adjuvant system) will be given intramuscularly at different intervals followed by a challenge with P. vivax infected mosquitoes. Safety, immunogenicity and efficacy parameters will be studied.

DETAILED DESCRIPTION:
This is a Phase 1/2a, non-randomized, open label, dose escalation study in healthy, malaria-naïve adults aged 18 to 55 years (inclusive). The vaccine will be administered with GlaxoSmithKline Biologicals' adjuvant system AS01B. This is a first-in-human study of VMP001; therefore the study design will incorporate a dose-escalation phase evaluating 15 µg, 30 µg, and 60 µg doses of VMP001 in 500 µL of AS01B. A total of 30 volunteers, divided into 3 groups (10 in each group), will receive 3 doses of the VMP001/AS01B vaccine. Group 1 will receive 15 µg of VMP001, Group 2 will receive 30 µg of VMP001, and Group 3 will receive 60 µg of VMP001 at each immunization. The dose of AS01B will be 500 µL for all groups. The first and second dose in each group will be separated by 28 days. The third dose in the three groups will be given at intervals scheduled to normalize the time to challenge between the last immunization and challenge. The second and third dose in Group 1 will be separated by 56 days, Group 2 by 42 days and Group 3 by 28 days. The challenge will occur 2 weeks following the third immunization. A group of 6-12 infectivity controls will begin participation in the study at the challenge stage. They will not receive any immunizations or placebos prior to challenge. All volunteers will receive a standard treatment regimen consisting of chloroquine and primaquine on the day that parasitemia is detected. Volunteers who do not become parasitemic will also begin the same treatment regimen on day 28 following the challenge (study day 126).

>

> Safety and immunogenicity will be evaluated during the study through the final study visit 6 months after challenge (study day 280).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet all of the following criteria may participate in this study:
* Healthy adults (male or non-pregnant, non-lactating female) 18 to 55 years of age (inclusive) at the time of enrollment
* If the subject is female, she must be of non-childbearing potential (either surgically sterilized or one year post-menopausal) or, if of childbearing potential, she must be capable of preventing pregnancy, have a negative pregnancy test at the time of each vaccination, and must agree to continue such precautions until completion of the last study visit.
* Free of significant health problems as established by medical history, laboratory and clinical examination before entering the study
* Duffy positive phenotype (homozygous or heterozygous)
* Normal (non-deficient) Glucose 6-phosphate dehydrogenase (G6PD) phenotype (range: 4.6 to 13.5 units/gm hemoglobin)
* Volunteers must have low cardiac risk factors according to the NHANES I criteria and a non-significant electrocardiogram (EKG)
* Available to participate and reachable by phone for duration of study (approximately 9 months)
* No plans to travel to outside the Washington, District of Columbia (DC) area up until treatment course has been completed (post challenge)
* No plans to travel to a malaria endemic area during the course of the study
* Written informed consent must be obtained from the subject before screening procedures
* Volunteers must score at least 80% correct on a 10 or 14 question multiple-choice quiz (control and immunization groups, respectively) that assesses their understanding of this study
* If a subject is active duty military he or she must obtain approval from his or her supervisor per Walter Reed Army Institute of Research (WRAIR) Policy 06-15

Exclusion Criteria:

* Subjects meeting any of the following criteria will be excluded from the study:
* Any history of malaria infection
* History of travel to P. vivax endemic areas in the last three months, and travel to Republic of Korea or China in the last 18 months
* Any history of receiving malaria vaccine or any licensed vaccine within 7 days prior to first immunization
* History of receipt of malaria prophylaxis during the previous 2 months or the use of any drugs with significant anti-malarial activity during the study period one month prior to challenge (for control volunteers). Examples include tetracycline, doxycycline, clindamycin, azithromycin or sulfa drugs
* Use of any investigational or non-registered drug or vaccine within 30 days preceding the first dose of study vaccine or planned use during the study period.
* Any history of allergic reaction or anaphylaxis to previous vaccination

Allergy to kanamycin, nickel, or imidazole

* Pregnant (positive β-HCG) or nursing at screening or plans to become pregnant or nurse from the time of enrollment until study completion.
* Allergy to antimalarial drugs or use of medications known to cause drug reactions with chloroquine and/or primaquine
* Significant (e.g. systemic) hypersensitivity reactions to mosquito bites (local hypersensitivity reactions at the site of mosquito bites are not an exclusion criterion)
* History of sickle cell disease
* History of psoriasis or porphyria
* History of splenectomy
* Any confirmed or suspected immunodeficiency, including HIV infection
* Administration of chronic (defined as more than 14 days) immunosuppressive drugs or other immune-modifying drugs within 6 months of immunization. For corticosteroids, this is defined as >20 mg/day prednisone or equivalent. -Inhaled and topical steroids are allowed
* A family history of congenital or hereditary immunodeficiency
* Acute or chronic, clinically significant, pulmonary, cardiovascular, hepatic, or renal functional abnormality, as determined by history, physical examination, and laboratory evaluation
* History of diabetes or hypertension even if well controlled on medication
* An abnormal baseline screening electrocardiogram (EKG) suggestive of cardiac disease as determined by a clinical investigator
* Chronic or active neurologic disease including seizure disorder and chronic migraine headaches
* Any abnormal baseline laboratory screening tests: Alanine Aminotransferase (ALT) above normal range, -Creatinine above normal range, Hemoglobin out of normal range, Platelet count out of normal range, Total white blood cell count out of normal range
* Hepatomegaly, right upper quadrant abdominal pain or tenderness
* Seropositive for HIV or hepatitis C virus, or HBsAg positive
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine or any planned administration during the study period
* Suspected or known current alcohol or drug abuse as determined from the medical history or by physical examination
* Any other significant finding that in the opinion of the investigator would increase the risk of having an adverse outcome from participating in this study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Bennett, MD, Principal Investigator — Division of Malaria Vaccine Development (DMVD), Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- Clinical Trials Center, Walter Reed Army Institute of Reserach, Silver Spring, Maryland, United States

REFERENCES:
- [Result] Bennett JW, Pybus BS, Yadava A, Tosh D, Sousa JC, McCarthy WF, Deye G, Melendez V, Ockenhouse CF. Primaquine failure and cytochrome P-450 2D6 in Plasmodium vivax malaria. N Engl J Med. 2013 Oct 3;369(14):1381-2. doi: 10.1056/NEJMc1301936. No abstract available. PMID 24088113
- [Derived] Kamau E, Bennett JW, Yadava A. Safety and Tolerability of Mosquito Bite-Induced Controlled Human Infection with Plasmodium vivax in Malaria-Naive Study Participants-Clinical Profile and Utility of Molecular Diagnostic Methods. J Infect Dis. 2022 Jan 5;225(1):146-156. doi: 10.1093/infdis/jiab332. PMID 34161579

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 41 patients were enrolled (30 vaccination group, 6 infectivity control group and 5 alternates) and received treatment at the Clinical Trials Center (CTC) at Walter Reed Army Institute of Research (WRAIR)
Groups:
- Cohort 1: 15 μg VMP001: 15ug VMP001 per vaccination on days -1 or 0, 28, and 84. P. vivax sporozoite challenge on day 98.
  VMP001: Plasmodium vivax malaria protein 001 (VMP001) with GlaxoSmithKline (GSK) Biologicals' Adjuvant System AS01B (Adjuvant Formulation)
  P. vivax sporozoite challenge: P. vivax sporozoite challenge
Period: Overall Study
Arm/Group | Cohort 1: 15 μg VMP001 | Cohort 2: 30 μg VMP001 | Cohort 3: 60 μg VMP001 | Control
Started | 10 | 10 | 10 | 6
Completed | 8 | 8 | 10 | 5
Not Completed | 2 | 2 | 0 | 1
Not completed — Lost to Follow-up | 2 | 0 | 0 | 1
Not completed — Relocated | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: 15 μg VMP001 | Cohort 2: 30 μg VMP001 | Cohort 3: 60 μg VMP001 | Control | Total
Number analyzed (Participants) | 10 | 10 | 10 | 6 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.1 (8.3) | 29.4 (8.2) | 28.7 (8.0) | 25.0 (7.2) | 30.1 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 4 | 3 | 13
  Male | 6 | 8 | 6 | 3 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 10 | 6 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 0 | 4
  White | 7 | 9 | 8 | 4 | 28
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 6 | 36

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Solicited Adverse Events Over a 7 Day Follow-up Period After Each Immunization (the Day of the Immunization and 6 Subsequent Days) During the Vaccination Phase
Description: Adverse events were evaluated for 7 days after each vaccination during the vaccine phase.
Time Frame: 7 days after immunization
Population: Control group was not included in the evaluation.
Measure: Number; unit: participants with AEs
Arm/Group | Cohort 1: 15 μg VMP001 | Cohort 2: 30 μg VMP001 | Cohort 3: 60 μg VMP001
Number analyzed (Participants) | 10 | 10 | 10
participants with AEs
  Solicited Local: Injection site erythema | 2 | 3 | 6
  Solicited Local: Injection site induration | 0 | 1 | 2
  Solicited Local: Injection site pain | 10 | 10 | 10
  Solicited Systemic: Diarrhea | 0 | 0 | 1
  Solicited Systemic: Nausea | 5 | 3 | 4
  Solicited Systemic: Vomiting | 2 | 0 | 2
  Solicited Systemic: Fatigue | 8 | 4 | 7
  Solicited Systemic: Pyrexia | 4 | 2 | 1
  Solicited Systemic: Arthralgia | 4 | 2 | 3
  Solicited Systemic: Myalgia | 4 | 4 | 7
  Solicited Systemic: Headache | 8 | 6 | 5

2. Primary Outcome: Occurrence of Unsolicited Adverse Events Over a 28 Day Follow-up Period After Each Immunization (the Day of the Immunization and 27 Subsequent Days) During the Vaccination Phase
Description: Adverse events were evaluated over a 28 day follow-up period after each vaccination during the vaccine phase
Time Frame: 28 days following immunization
Population: Control group was not included in this evaluation.
Measure: Number; unit: participants with AEs
Arm/Group | Cohort 1: 15 μg VMP001 | Cohort 2: 30 μg VMP001 | Cohort 3: 60 μg VMP001
Number analyzed (Participants) | 10 | 10 | 10
participants with AEs
  Ear discomfort | 1 | 0 | 0
  Abdominal discomfort | 1 | 0 | 0
  Abdominal pain | 0 | 0 | 1
  Feces discolored | 0 | 0 | 1
  Food poisoning | 1 | 0 | 0
  Nausea | 1 | 0 | 0
  Toothache | 2 | 0 | 0
  Axillary pain | 0 | 1 | 0
  Chills | 5 | 5 | 7
  Feeling hot | 5 | 6 | 7
  Injection site erythema | 0 | 0 | 1
  Injection site pruritus | 0 | 0 | 1
  Injection site swelling | 0 | 2 | 3
  Injection site warmth | 0 | 1 | 2
  Malaise | 3 | 5 | 7
  Hypertransaminasaemia | 1 | 2 | 1
  Seasonal allergy | 1 | 0 | 1
  Nasopharyngitis | 1 | 0 | 0
  Upper respiratory tract infection | 2 | 0 | 2
  Contusion | 0 | 0 | 1
  Excoriation | 0 | 0 | 1
  Postprocedural discomfort | 0 | 1 | 0
  Posttraumatic pain | 0 | 0 | 1
  Scratch | 0 | 0 | 1
  Skin laceration | 0 | 0 | 2
  Haemoglobin decreased | 0 | 1 | 1
  Platelet count decreased | 0 | 1 | 1
  Gout | 1 | 0 | 0
  Back pain | 0 | 1 | 1
  Muscle spasms | 1 | 0 | 0
  Musculoskeletal discomfort | 1 | 0 | 1
  Myalgia | 1 | 0 | 0
  Pain in extremity | 2 | 0 | 2
  Dizziness | 1 | 0 | 1
  Headache | 1 | 0 | 0
  Sinus headache | 0 | 0 | 1
  Nasal Congestion | 0 | 0 | 1
  Cold sweat | 2 | 4 | 2
  Dermatitis contact | 0 | 1 | 0
  Erythema | 0 | 1 | 0
  Hypertension | 1 | 0 | 0

3. Primary Outcome: Occurrence of Serious Adverse Events at Any Time During the Study Period (Enrollment to Final Follow up Visit)
Description: Occurrence of serious adverse events at any time during the approximately 463 day study period
Time Frame: up to 463 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 15 μg VMP001 | Cohort 2: 30 μg VMP001 | Cohort 3: 60 μg VMP001 | Control
Number analyzed (Participants) | 10 | 10 | 10 | 6
Participants
  Not Related to study drug - Breast cancer (left) | 1 | 0 | 0 | 0
  Related to study drug | 0 | 0 | 0 | 0
  Patients without SAE | 9 | 10 | 10 | 6

4. Secondary Outcome: Time to Parasitemia for Immunogenicity Population
Description: Subjects were ranked according to time of onset of parasitemia and a non-parametric rankorder statistical test (eg, Log-Rank or Mann-Whitney) was performed to evaluate delays in parasitemia induced by vaccination. Cox Proportional Hazards model was used to calculate days to parasitemia and Kaplan-Meier plots were used to display time to first positive malaria blood smear.
  Hazard Ratio (HR). Time starts once subject has received t infectious bites. Time stops when subject has first positive blood smear. If subject does not become parasitemic then time stops the day he/she begins anti-malarial therapy.
Time Frame: 280 day (during the study through 6 months aftr challenge)
Population: Drop-outs prior to vaccination were not included in the analysis
Measure: Mean (Standard Error); unit: days
Arm/Group | Cohort 1: 15 μg VMP001 | Cohort 2: 30 μg VMP001 | Cohort 3: 60 μg VMP001
Number analyzed (Participants) | 9 | 8 | 10
days | 0.137 (2.025) | 0.073 (2.106) | 0.042 (2.154)

5. Secondary Outcome: Geometric Mean of Anti-VMP001 Antibody Titers in Serum Per Immunogenicity Population
Description: Anti-VMP001 antibody concentrations were measured and summarized by geometric mean titers (GMT) with 95% confidence interval (CI). Peak responses were compared by performing Student's t-test on data normalized by log transformation to ascertain the presence or absence of significant dose response differences. ELISA Units (EU) were converted to log10 values for calculations and statistical comparison of geometric means. Units that were reported as '>50' were converted to '1'.
Time Frame: study duration
Population: Immunogenicity population
Measure: Mean (95% Confidence Interval); unit: Geometric Mean Titer of European Units
Arm/Group | Cohort 1: 15 μg VMP001 | Cohort 2: 30 μg VMP001 | Cohort 3: 60 μg VMP001
Number analyzed (Participants) | 10 | 10 | 10
Geometric Mean Titer of European Units
  Pre-vaccination | 1 [1 to 1] | 1.5 [0.6 to 3.76] | 3.09 [0.56 to 17.05]
  2wks post first vaccination | 151.39 [31.62 to 724.71] | 526.18 [194.01 to 1427.06] | 836.68 [147.84 to 4735.05]
  Day of second vaccination: number analyzed (Participants) | 10 | 9 | 10
  Day of second vaccination | 281.79 [53.6 to 1481.36] | 1175.41 [391.29 to 3530.89] | 1711.63 [685.48 to 4273.89]
  2wks post second vaccination: number analyzed (Participants) | 10 | 9 | 10
  2wks post second vaccination | 21862.22 [10775.91 to 44354.18] | 74608.62 [51309.78 to 108487.04] | 61711.8 [33584.06 to 113397.42]
  Day of third vaccination: number analyzed (Participants) | 10 | 9 | 10
  Day of third vaccination | 9921.61 [5707.48 to 17247.25] | 28498.43 [18863.52 to 43054.55] | 36405.66 [19839.55 to 66804.57]
  2wks post third vaccination: number analyzed (Participants) | 10 | 8 | 10
  2wks post third vaccination | 59883.77 [38915.79 to 92149.38] | 68730.4 [48391.1 to 97618.54] | 41879.99 [22137.62 to 79228.66]
  4wks post challenge: number analyzed (Participants) | 9 | 8 | 10
  4wks post challenge | 54843.38 [34557.05 to 87038.59] | 56472.17 [38216.28 to 83448.88] | 32178.39 [17659.05 to 58635.6]
  6months post challenge: number analyzed (Participants) | 8 | 8 | 10
  6months post challenge | 10860.7 [5151.41 to 22897.6] | 12519.16 [5950.55 to 26338.62] | 5500.73 [2751.67 to 10996.23]

6. Secondary Outcome: Geometric Mean of Anti-VMP001 Anti-body Titers in Serum Per Efficacy Population
Description: as for outcome 5
Time Frame: study duration
Population: Efficacy population
Measure: Mean (95% Confidence Interval); unit: Geometric Mean Titier of European Units
Arm/Group | Cohort 1: 15 μg VMP001 | Cohort 2: 30 μg VMP001 | Cohort 3: 60 μg VMP001
Number analyzed (Participants) | 9 | 8 | 10
Geometric Mean Titier of European Units
  Pre-vaccination | 1 [1 to 1] | 1 [1 to 1] | 3.09 [0.56 to 17.05]
  2wks post first vaccination | 133.72 [23.1 to 774] | 750.38 [251.51 to 2238.74] | 836.68 [147.84 to 4735.05]
  Day of second vaccination | 244.35 [38.22 to 1562.29] | 1450.22 [460.04 to 4571.68] | 1711.63 [685.48 to 4273.89]
  2wks post second vaccination | 20161.18 [9253.42 to 43926.79] | 81143.72 [55905.91 to 117774.72] | 61711.8 [33584.06 to 113397.42]
  Day of third vaccination | 9053.32 [5047.3 to 16238.9] | 31071.01 [20413.38 to 47292.88] | 36405.66 [19839.55 to 66804.57]
  2wks post third vaccination | 61203.48 [37570.19 to 99703.16] | 68730.4 [48391.1 to 97618.54] | 41879.99 [22137.62 to 79228.66]
  4wks post challenge | 54843.38 [34557.05 to 87038.59] | 56472.17 [38216.28 to 83448.88] | 32178.39 [17659.05 to 58635.6]
  6mths post challenge | 10860.7 [5151.41 to 22897.6] | 12519.16 [5950.55 to 26338.62] | 5500.73 [2751.67 to 10996.23]

ADVERSE EVENTS:
Groups:
- Cohort 1: 15 μg VMP001: 01
- Cohort 2: 30 μg VMP001: 02
- Cohort 3: 60 μg VMP001: 03
- Cohort 4: Control: 04
Arm/Group | Cohort 1: 15 μg VMP001 | Cohort 2: 30 μg VMP001 | Cohort 3: 60 μg VMP001 | Cohort 4: Control
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8 | 0/10 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/8 | 0/10 | 1/6
Other Adverse Events (participants affected / at risk) | 9/9 | 8/8 | 10/10 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: 15 μg VMP001 (N=9) | Cohort 2: 30 μg VMP001 (N=8) | Cohort 3: 60 μg VMP001 (N=10) | Cohort 4: Control (N=6)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: 15 μg VMP001 (N=9) | Cohort 2: 30 μg VMP001 (N=8) | Cohort 3: 60 μg VMP001 (N=10) | Cohort 4: Control (N=6)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1) | 7 (9) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (3) | 2 (3)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 6 (7) | 9 (10) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 4 (5) | 6 (7) | 7 (7) | 0 (0)
Fatigue (General disorders) | 5 (6) | 6 (6) | 10 (11) | 5 (9)
Feeling hot (General disorders) | 1 (1) | 1 (1) | 3 (3) | 4 (4)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 1 (2) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 5 (7) | 6 (6) | 5 (8) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 2 (4) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3) | 3 (3) | 2 (2)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5) | 5 (5) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 4 (5) | 9 (9) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (7) | 5 (7) | 8 (9) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (4) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 2 (4) | 2 (2) | 1 (1) | 1 (2)
Paraesthesia (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (3) | 4 (5) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No